CLINICAL TRIAL: NCT04541758
Title: Comparing the Efficacy of Conservative Treatment With Minimally Invasive Surgery in the Treatment of 2-4 Displaced Rib Fractures:A Prospective Randomized Controlled Study
Brief Title: Comparing the Efficacy of Conservative Treatment With Minimally Invasive Surgery in the Treatment of Rib Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Li Yang, Principal Investigator, Shanghai 6th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ynlc201908
Record Dates: First submitted 2020-08-15; First posted 2020-09-09 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Chest Trauma; Rib Fractures; Surgery--Complications
Keywords: rib fractrue;surgical treatment;Rapid recovery
MeSH Terms: conditions — Thoracic Injuries; Rib Fractures | interventions — Surgical Procedures, Operative; Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgical treatment (Experimental): Minimally invasive internal fixation under spontaneous respiratory anesthesia and analgesic treatment and chest strap fixation
  Interventions: Procedure: surgical treatment; Procedure: Conservative treatment
- Conservative treatment (Experimental): analgesic treatment and chest strap fixation
  Interventions: Procedure: Conservative treatment

INTERVENTIONS:
Procedure: surgical treatment — surgical treatment and Conservative treatment
  Arms: surgical treatment
Procedure: Conservative treatment — Conservative treatment

SUMMARY:
Open, randomized, parallel controlled prospective clinical study design was used in this study.Subjects were patients with 2-4 displaced non-flail rib fractures.Operation group (Group 1) : minimally invasive internal fixation operation group under spontaneous breathing anesthesia.In the operation group of minimally invasive internal fixation under autonomic respiratory anesthesia, the fracture was determined preoperatively by chest CT+ three-dimensional reconstruction of the ribs, and the optimal incision location was determined. The fracture was exposed through as many small incisions as possible, and fixed with titanium plate or clon-type plate. During the operation, the autonomic respiratory anesthesia and paraviral nerve block technology was adopted.In the conservative group (group 2), routine treatment measures such as analgesia and chest strap fixed were adopted.The purpose of this study was to evaluate the safety, feasibility, and efficacy of minimally invasive and conservative treatment for rib fractures with different Numbers of displaced ends.

DETAILED DESCRIPTION:
An open, randomized, parallel controlled prospective clinical study design type was used in this study. Subjects were patients with two to four displaced non-flail chest fractures of the ribs. Operation group (Group 1) : minimally invasive internal fixation operation group under spontaneous breathing anesthesia. In the operation group of minimally invasive internal fixation under autonomic respiratory anesthesia, the fracture was determined preoperatively by chest CT+ three-dimensional reconstruction of the ribs, and the optimal incision location was determined. The fracture was exposed through as many small incisions as possible, and fixed with titanium plate or clon-type plate. During the operation, the autonomic respiratory anesthesia and paraviral nerve block technology was adopted. In the conservative group (group 2), routine treatment measures such as analgesia, hemostasis and chest band fixation were adopted. The effects of the two treatments on lung function, pain index, complications and QoL were evaluated. It provides theoretical basis for the treatment of rib fracture

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral thoracic trauma, fractured ends of rib fractures displaced 2-4 places
2. Displaced fracture（CT image shows double displacement of bone cortex） located in the 3rd to 10th rib
3. The number of broken ends of displaced fractures is greater than that of undisplaced fractures
4. The length of time from injury to hospitalization <24 hours
5. Age range（18-70）
6. ASA grade I-II
7. BMI < 30
8. Preoperative partial arterial oxygen pressure >60mmHg, partial arterial carbon dioxide pressure <50mmHg

Exclusion Criteria:

1. Difficult airway
2. History of esophageal reflux
3. Myasthenia gravis
4. Abnormal coagulation system
5. History of gastrointestinal ulcer or bleeding
6. History of anaesthesia related drug allergy

A history of asthma or chronic obstructive emphysema

8. Women during pregnancy

9. Flail chest

10. Combined with severe craniocerebral trauma and external abdominal injuries

11. Recent use of clopidogrel, warfarin and aspirin seriously affects blood clotting

12. Self-administered analgesics after injury

13.Massive hemopneumothorax requires emergency surgery

14. Patients who cannot tolerate surgery

-

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2023-06-10 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage improvement of lung function FEV1(Forced expiratory volume in one second) | FEV1%(One week after treatment)-FEV1%(Admitted)
  FEV1(Forced expiratory volume in one second)，FEV1% ：percentage of the expected value

SECONDARY OUTCOMES:
Percentage improvement of lung function FVC | FVC%(One week after treatment)-FVC%(Admitted)
  FVC（forced vital capacity），FVC%：percentage of the expected value
Percentage improvement of lung function PEF | PEF%(One week after treatment)-PEF%(Admitted)
  PEF（peak expiratory flow ），PEF%：percentage of the expected value
Pain index | Admitted；One week after treatment；One month after treatment;Three month after treatment;Half a year;One year
  visual analogue scale，VAS（0-10）0：no pain；10：severe pain
Pleural effusion | Admitted；One week after treatment；One month after treatment;Three month after treatment;Half a year;One year
  Measured by chest CT
Mortality rate | Admitted；One week after treatment；One month after treatment;Three month after treatment;Half a year;One year
  Deaths associated with this study
Length of hospital stay | Admitted；One week after treatment；One month after treatment;Three month after treatment;Half a year;One year
  Length of hospital stay
Cost of treatment | One year
  Sum of all treatment costs
Chronic pain | Three month after treatment;Half a year;One year
  Pain lasting more than three months（It is suggested in the related article that pain lasting more than 3 months is chronic pain）visual analogue scale，VAS（0-10）0：no pain；10：severe pain
Quality of Life score | One week after treatment；One month after treatment;Three month after treatment;Half a year;One year
  The Barthel index of ADL
Time to resume routine work | One week after treatment；One month after treatment;Three month after treatment;Half a year;One year
  Time to resume routine work
Duration of analgesic medication | intraoperative；One week after treatment；One month after treatment;Three month after treatment;Half a year;One year
  Duration of analgesic medication

CONTACTS AND LOCATIONS:
Overall Officials: Yi Yang, PHD, Study Director — Shanghai 6th People's Hospital; Zongli Gao, PHD, Study Chair — Shanghai 6th People's Hospital; Yonghong Zhao, PHD, Study Chair — Shanghai 6th People's Hospital; Weiming Wu, PHD, Study Chair — Shanghai 6th People's Hospital; Weigang Zhao, PHD, Study Chair — Shanghai 6th People's Hospital; Tiancheng Zhao, PHD, Study Chair — Shanghai 6th People's Hospital; Xiang Guo, PHD, Study Chair — Shanghai 6th People's Hospital; Lei Wang, PHD, Study Chair — Shanghai 6th People's Hospital; Weiwei He, PHD, Study Chair — Shanghai 6th People's Hospital

IPD SHARING:
Plan to Share IPD: No
The data will not be Shared with other researchers